CLINICAL TRIAL: NCT01237561
Title: Translating The GOLD COPD Guidelines Into Primary Care Practice
Acronym: LungAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Donna R. Parker, Associate Professor of Family Med & Epidemiology, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08-19; R01HL093090 (NIH)
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; COPD Guidelines; Patient Activation; Lung Age
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- spirometry, patient activation tool (Experimental): * Receive Portable Spirometer
  * Spirometry training of staff
  * Provide clinician with web-based COPD interactive guideline tool
  * Provide clinician with patient activation tool
  * Train clinicians (tools, integration into workflow)
  * Academic Detailing
  Interventions: Other: provider support tools plus spirometer
- Usual Care (No Intervention): Spirometer and spirometry training of staff

INTERVENTIONS:
Other: provider support tools plus spirometer — Patient Activation Tool, Provider Web-based decision support tool, academic detailing
  Other Names: Determine the effectiveness of tools developed in improving guideline implementation and adherence.
  Arms: spirometry, patient activation tool

SUMMARY:
This project will evaluate the translation of the Gold (the Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease) COPD guidelines into primary care practice. During phase I, a needs assessment will evaluate barriers and facilitators to implementation of COPD guidelines into clinical practice through focus groups of primary care patients and providers. Using formative evaluation and feedback from the focus groups, three tools will be developed, refined and pilot tested. The effectiveness of the materials developed in phase I will be tested in phase II (a randomized clinical trial conducted with one year of intervention within non-academic primary care practices) regarding physician performance of COPD guideline implementation and improvement in the clinically relevant outcomes (appropriate screening, diagnosis and management of COPD) compared to usual care.

DETAILED DESCRIPTION:
This project will evaluate the translation of the GOLD (the Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease) COPD guidelines into primary care practice. This study is based upon the premise that an informed, activated patient will interact with a prepared, proactive team to improve appropriate COPD screening, diagnosis and management. During phase I, a needs assessment will evaluate barriers and facilitators to implementation of COPD guidelines into clinical practice through focus groups of primary care patients and providers. Using formative evaluation and feedback from the focus groups, three tools will be developed, refined and pilot tested. These include: a computerized patient activation tool that will be used by the patient either in the waiting room or in the examination room; a web-based, interactive COPD guidelines tool to be used by primary care providers as a decision support tool at the point of care and a COPD patient education toolbox to be used by the practice team. During phase II, a block, randomized design cluster trial will be performed with one year of intervention within non-academic primary care practices (30 practices) throughout the state of Rhode Island and southeastern MA. The effectiveness of the materials developed in phase I will be tested in phase II regarding physician performance of COPD guideline implementation and the improvement in the clinically relevant outcomes (appropriate screening, diagnosis and management of COPD) compared to usual care. The investigators will also examine the use of a patient activation tool -'MyLungAge' to prompt patients to talk with their health care provider regarding their lung health and risk for COPD. Products for dissemination from this grant will include the results of the focus groups barriers and facilitators to implementation and adherence to COPD guidelines, a computerized data collection module for quality of care assessment regarding COPD guidelines, a refined computerized patient activation tool, an enhanced web-based COPD interactive guideline tool, tailored academic detailing materials, and the results of the randomized clinical trial on the effectiveness of these tools to improve COPD guideline adherence in primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients 40 years or older
* Seen at least once in the past 2 years (active patients) by their PCP
* And/or 40 years of age and less than 81 years of age who smoke.

Exclusion Criteria:

* < 40 years of age

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3593 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-10-25 (Actual); Study Completion 2013-10-25 (Actual)

PRIMARY OUTCOMES:
Adherence to COPD guidelines | Twelve months post intervention
  An adherence tool will be developed and reviewed by an expert panel. They will review the suggested criterion and make recommendations regarding an item's status on the tool. The panel may also suggest additional criteria for inclusion in the tool. The tool will be modified based on expert consensus. Once the tool is finalized, a detailed algorithm will be developed for scoring the primary care practice data which will include an adherence score for each visit and an overall adherence score and will be piloted the first 2 months of chart review.

SECONDARY OUTCOMES:
patient activation | Baseline and 12 months post intervention
  A patient activation measure (PAM) developed by Hibbard et al. will be used to assess a patient's knowledge, skills and behaviors necessary to create an activated patient for managing their own health care. The patient activation tool will also measure other co-morbidities and will be assessed during a telephone survey at baseline and on a subsample 12 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Parker, Sc.D., Principal Investigator — MHRhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

REFERENCES:
- [Derived] Parker DR, Eaton CB, Ahern DK, Roberts MB, Rafferty C, Goldman RE, McCool FD, Wroblewski J. The study design and rationale of the randomized controlled trial: translating COPD guidelines into primary care practice. BMC Fam Pract. 2013 May 6;14:56. doi: 10.1186/1471-2296-14-56. PMID 23641803